CLINICAL TRIAL: NCT05781282
Title: Pulmonary Vein Imaging by ICE After Atrial Fibrillation Ablation to Predict Recurrences
Brief Title: Pulmonary Vein (PV) Imaging by Intracardiac Echography (ICE) After Ablation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Bencardino Gianluigi, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 3747
Record Dates: First submitted 2023-03-01; First posted 2023-03-23 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Atrial Fibrillation Recurrent

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Atrial fibrillation ablation — Pulmonary vein deconnection. PV antra visualization by ICE

SUMMARY:
To test the hypothesis that structural changes documented by ICE after pulmonary vein deconnection by RF can predict AF recurrences

DETAILED DESCRIPTION:
Patient undergoing first RF ablation for sympomatic paroxysmal atrial fibrillation will be enrolled. ICE visualization of PV antra before and after PV deconnection (electrophysiological endpoint). Changes in echogenicity as documented by ICE will be evaluated by a dedicated software and correlated to long term recurrences

ELIGIBILITY:
Inclusion Criteria:

* Atrial fibrillation ablation candidates

Exclusion Criteria:

* Previous catheter ablation
* Persistent atrial fibrillation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation recurrences | 12 months
  Recurrences of atrial fibrillation at 12 months follow up despite pulmonary vein deconnection

CONTACTS AND LOCATIONS:
Overall Officials: Gianluigi Bencardino, Dr, Principal Investigator — Fondazione Policlinico Agostino Gemelli Roma IRCCS
Locations (1):
- Fondazione Policlinico Agostino Gemelli Roma IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Leo M, De Maria GL, Briosa E Gala A, Pope M, Banerjee A, Kelion A, Pedersen M, Rajappan K, Ginks M, Bashir Y, Hunter RJ, Betts T. INtra-procedural ultraSound Imaging for DEtermination of atrial wall thickness and acute tissue changes after isolation of the pulmonary veins with radiofrequency, cryoballoon or laser balloon energy: the INSIDE PVs study. Int J Cardiovasc Imaging. 2021 Dec;37(12):3525-3535. doi: 10.1007/s10554-021-02417-7. Epub 2021 Sep 23. PMID 34554367